CLINICAL TRIAL: NCT04196985
Title: Comparison Between 18F-FDG PET/CT and 18F-FDG PET/MRI in Detecting Locoregional Recurrence 3 Months After Chemoradiation Therapy (CRT) in Head and Neck Squamous Cell Carcinoma (SCC)
Brief Title: 18F-FDG PET/CT Versus 18F-FDG PET/MRI in Detecting Locoregional Recurrence 3 Months After CRT in Head and Neck SCC
Acronym: HENEPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HENEPET
Record Dates: First submitted 2019-11-20; First posted 2019-12-12 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: PET-imaging; local recurrence; PET/MRI; chemoradiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HNSCC (Experimental): Patients who have histologically confirmed HNSCC and have received CRT for it
  Interventions: Diagnostic Test: PET/MRI; Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/MRI — each patient will perform PET/CT and PET/MRI scans in two different days within the interval of less than 2 weeks receiving two different FDG injections. Administered FDG activity for each PET scan will be 4 MBq/Kg up to a maximum of 400 MBq.
Diagnostic Test: PET/CT — each patient will perform PET/CT and PET/MRI scans in two different days within the interval of less than 2 weeks receiving two different FDG injections. Administered FDG activity for each PET scan will be 4 MBq/Kg up to a maximum of 400 MBq.

SUMMARY:
Comparing FDG PET/CT and FDG PET/MRI in the diagnostic accuracy of detecting local recurrence 12 weeks after the end of CRT in head and neck squamous cell carcinoma patients. Forty patients aged more than 18 years who have a histologically confirmed HNSCC and have received chemoradiation therapy will be recruited for the study. The patients will be scanned with both PET/CT and PET/MRI 12 weeks after the end of CRT.

DETAILED DESCRIPTION:
Since recurrence of HNSCC occurs in up to 50 percent of cases in the first two years following treatments and the recurrent diseases are less responsive to new treatments, detecting local/regional recurrence at an earlier time is crucial in order to provide salvage treatments. The primary objective of this prospective study is to compare the diagnostic accuracy of FDG PET/CT to FDG PET/MRI in the detection of local recurrence 12 weeks after the end of chemoradiation treatment in HNSCC patients. The hypothesis is that PET/MRI might be able to diagnose locoregional recurrence earlier and more accurately which would lead to a better outcome for the patient. If it is proven correct, it would be possible to optimize the use of PET/MRI imaging on selected patients who are likely to benefit clearly from the use of that modality.

Forty patients aged more than 18 years who have a histologically confirmed HNSCC and have received chemoradiation therapy will be recruited for the study. The patients will be scanned with both FDG-PET/CT and FDG-PET/MRI 12 weeks after the end of CRT.

All study participants will be consented, and the estimated time for completing the PET scans of 40 patients will take 12 to 15 months. The results will be reported in international peer-reviewed high-impact journals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Language spoken: Finnish or Swedish
* Diagnosis: Histologically confirmed HNSCC
* Chemoradiotherapy treatment with curative intent to the primary tumor and/or neck LN metastasis that has ended 12+- 4 weeks before the PET scan.
* Clinical stage: Stage I-II at least 20 patients, Stage III-IV at least 20 patients
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient has to have signed the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Uncontrolled serious infection
* Contraindications for MRI (cardiac pacemaker, intracranial clips etc., allergic reaction to contrast agent)
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | 12 weeks after chemoradiotherapy
  local recurrence detected with PET/TT vs. with PET/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Kemppainen, MD PhD, Principal Investigator — Turku University Hospital PET Centre
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided